CLINICAL TRIAL: NCT07190885
Title: A Pharmacokinetic Study of YN001 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Inno Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YN001-103
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YN001 (Experimental): Approximately 24 healthy male and female volunteers (18-65 years) will receive a single dose of YN001. Participants will be assigned to one of two dose cohorts: Cohort 1 - 20 mg (n=12) or Cohort 2 - 40 mg (n=12)
  Interventions: Drug: YN001

INTERVENTIONS:
Drug: YN001 — YN001 administered via intravenous infusion. Participants will receive either 20 mg (Cohort 1) or 40 mg (Cohort 2).

SUMMARY:
This is a Phase 1, single-center, open-label study designed to evaluate the pharmacokinetics (PK), safety, and immunogenicity following a single dose administration in healthy adult volunteers.

DETAILED DESCRIPTION:
This will be a single center, open-label, single dose study in Healthy volunteers.

A total of approximately 24 healthy male and female participants will be enrolled into two dose groups (12 participants per dose group).

The study will consist of a maximum 27-day screening period, a baseline period (Day -1), a treatment period (Day 1), a follow up period (Day 2-15). After completion of relevant assessments on Day 8, participants will be followed for an additional 7 days and will have a completion visit conducted via phone call on Day 15.

The study is designed to refine PK profile of YN001 in Australian healthy volunteers to support further clinical development of YN001.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Healthy male and female adults aged from 18 to 65 years of age (inclusive) at time of Screening, and in good health as determined by no clinically significant (as judged by the PI/delegate) past medical history, physical examination, and vital signs, electrocardiogram (ECG), and laboratory tests at Screening and Baseline (Day -1).
3. Vital signs (systolic and diastolic blood pressure and pulse rate) measurements within the below ranges at Screening and Baseline (Day -1):

   * tympanic body temperature between 35.5-37.7 °C
   * systolic blood pressure, 90-140 mm Hg (inclusive)
   * diastolic blood pressure, 40-95 mm Hg (inclusive)
   * pulse rate, 40-100 bpm (inclusive)
4. Weigh at least 50 kg and have a body mass index (BMI) within the range of 18-32 kg/m2 at Screening and Baseline (Day -1).
5. Meets contraception requirements.
6. Willing and able to comply with the study requirements and restrictions.

Exclusion Criteria:

1. Received an investigational agent within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
2. Use of any prescription drugs, over the counter (OTC) medication, herbal supplements, dietary supplements (vitamins included), any type of vaccine within two weeks prior to the study drug administration, unless deemed acceptable by the Principal Investigator (or delegate) and agreement with the Sponsor.
3. Fasting triglyceride concentration >2.8 mmol/L at Screening or Baseline (Day -1).
4. A history of clinically significant ECG abnormalities, or any ECG abnormalities at Screening or Baseline (Day -1).
5. Pregnant or nursing (lactating) women.
6. Average use of more than 5 cigarettes or equivalent nicotine containing products per week and/or unwilling to abstain from such products 7 days prior to study administration through until Day 15. Positive urine cotinine test at Baseline (Day -1); repeat testing may be permitted at PI/delegate discretion.
7. History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by positive results for alcohol or drugs conducted at Screening and/or Baseline (Day -1). Alcohol abuse is defined as consumption of 14 or more standard drinks per week (where 1 unit = 375 mL of beer [3.5% alc/vol], 30 mL of 40% spirit or a 100 mL glass of wine [13%]). Any THC-containing products should not be used at least 7 days prior to Screening through until completion of Day 15.
8. A positive hepatitis B surface antigen (HBsAg), or positive hepatitis C virus (HCV) or human immunodeficiency virus (HIV) test result at Screening.
9. History of myopathy/myalgia, or susceptible to myopathy/rhabdomyolysis (e.g., hypothyroidism, family history of hereditary myopathy, previous muscle toxicity with HMG CoA reductase inhibitors or fibrates).
10. Multiple drug allergies, or history of allergic reactions to study drug or any components of the study drug.
11. Donation or loss of more than 400 ml of blood within 3 months prior to study drug administration.
12. Plasma donation (> 100 ml) within 60 days prior to first dosing.
13. Hemoglobin levels below 120 g/L at Screening or Baseline (Day -1).
14. Recent (within the last 3 years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
15. Recent (within the last 3 years) and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated), or cardiac dysfunction or myocardial infarction.
16. History of significant food allergies (e.g. anaphylactic reactions). Mild (non-anaphylactic, hypersensitivity) food allergies such as lactose intolerance/glucose intolerance are permitted.
17. Any surgical or medical condition which might significantly alter the distribution, metabolism, or excretion of drugs, or which may jeopardize the participant in case of participation in the study. The Investigator should make this determination in consideration of the participant's medical history and/or clinical or laboratory evidence of any of the following:

    1. Inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding in the last 6 months.
    2. Pancreatic injury or pancreatitis in the last 6 months.
    3. Liver disease or liver injury as indicated by abnormal liver function tests at Screening or Baseline (Day -1) such as SGOT (AST), SGPT (ALT), GGT, alkaline phosphatase (ALP), or total bilirubin. The Investigator should be guided by the following criteria:

       • Any single parameter of ALT, AST, GGT, ALP, or total bilirubin must not exceed 1.5 x upper limit of normal (ULN).
    4. History or presence of impaired renal function as indicated by abnormal creatinine and/or urea values (e.g., eGFR<90 mL/min/1.73 m2 (calculated by CKD-EPI equation), or abnormal urinary constituents (e.g., albuminuria), deemed clinically significant by the PI/delegate at Screening or Baseline (Day -1).
    5. Evidence of urinary obstruction or difficulty in voiding at Screening.
18. Significant illness resolved within two weeks prior to dosing, which may affect the study drug administration and safety assessments in the opinion of the PI/delegate.
19. Any other medical condition or social circumstance, which in the opinion of the PI/delegate would impede compliance with or hinder completion of the study or otherwise deem the participant unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
To evaluate the maximum plasma concentration (Cmax) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be measured to determine Cmax.
To evaluate the time to reach maximum plasma concentration (Tmax) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be measured to determine Tmax.
To evaluate the area under the concentration-time curve from time 0 to last measurable concentration (AUC0-t) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be used to calculate AUC0-t.
To evaluate the area under the concentration-time curve extrapolated to infinity (AUCinf) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be used to calculate AUCinf.
To evaluate the terminal elimination rate constant (λz) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be used to estimate λz.
To evaluate the plasma half-life (T1/2) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be used to calculate T1/2.
To evaluate the clearance (CL) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be used to calculate clearance.
To evaluate the volume of distribution (Vd) of YN001 | From pre-dose (Day 1) through 120 hours post-dose (Day 6).
  Plasma concentration values will be used to calculate volume of distribution.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 15 days
  Number and percentage of participants with treatment-emergent AEs and SAEs as assessed by CTCAE v5.0.
Incidence of Anti-PEG Antibodies (APA) | From pre-dose (D1),Day 5, and Day 8.
  Characterization of anti-PEG antibodies, including the detection rate of pre-existing APAs and the emergence or boosting of treatment-induced APAs.
Change from Baseline in Laboratory Parameters | Up to 15 days
  Number and percentage of participants with clinically significant abnormalities in hematology, chemistry, or urinalysis.
Change from Baseline in Electrocardiogram (ECG) Parameters | Up to 15 days
  Number and percentage of participants with clinically significant ECG abnormalities after resting supine ≥5 minutes.
Change from Baseline in Vital Signs | Up to 15 days
  Number and percentage of participants with clinically significant abnormalities in systolic and diastolic blood pressure, pulse, and body temperature.
Change from Baseline in Physical Examination Findings | Up to 15 days
  Number and percentage of participants with clinically significant abnormalities in physical exam findings.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No